CLINICAL TRIAL: NCT03274349
Title: Influence of Whole Body Electromyostimulation and Nutritional Therapy for Patients With Esophageal and Bronchial Carcinoma in Curative and Palliative Treatment
Brief Title: Whole Body Electromyostimulation and Nutritional Therapy for Patients With Esophageal and Bronchial Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EMS Nutr ÖsoBroCA
Record Dates: First submitted 2017-05-30; First posted 2017-09-06 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cancer of Esophagus; Cancer, Lung
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, controlled pilot study
Who Masked: Outcomes Assessor
Masking Description: The patients will be coded by a consecutive numbering. Data will be saved only with this number. Access to the data will only be provided to authorized personnel (study nurses) and will be retained in inaccessable and locked rooms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Group of patients receiving individualized protein-rich nutritional therapy without exercise, 12 weeks intervention per patient
  Interventions: Procedure: protein-rich nutrition therapy
- EMS-group (Experimental): Group of patients receiving individualized protein-rich nutritional therapy with personalized whole body electromyostimulation exercise, 12 weeks intervention per patient
  Interventions: Procedure: whole body electromyostimulation exercise; Procedure: protein-rich nutrition therapy

INTERVENTIONS:
Procedure: whole body electromyostimulation exercise — whole body electromyostimulation exercise training twice a week for 20 min each, bipolar, 85 Hz, intermittent pulse/pause, pulse width 350 µsec
  Arms: EMS-group
Procedure: protein-rich nutrition therapy — protein-rich nutrition therapy with an objective of reaching 1,2 to 1,5 g protein/kg body weight and day

SUMMARY:
The objective or the trial is to study the influence of a combined therapy involving protein-rich individualized nutritional therapy and highly effective muscle training via personalized whole-body electromyostimulation exercise on muscle mass, muscle functionality, physical capability, fatigue and quality of life in patients with esophageal and bronchial carcinoma in advanced or metastatic stage.

DETAILED DESCRIPTION:
Tumor specific and inflammation promoting mediators lead to a loss of appetite, to systemic inflammation processes and to metabolic and hormonal changes including anabolic resistance. Consequences hereof are a decreased food uptake, a deteriorated nutrient utilization and a loss of muscles and/or fat leading to cancer cachexia. In addition, an accelerated muscle wasting can be a side effect of the oncologic therapy promoting cancer cachexia even further. The advancing muscle loss induces diminishing physical capability, a decreased tolerance of oncological therapy, functional losses even reaching loss of independence and a worsened prognosis.

The purpose of this study is to establish an innovative combined therapy involving protein-rich nutritional therapy and highly effective muscle training by personalized whole-body electromyostimulation (WB-EMS) exercise to improve muscle mass, functionality and strength of esophageal and bronchial carcinoma patients in advanced stage. An increase in muscle mass and strength leads to an increase in physical activity, physical capability as well as tolerance to and applicability of tumor therapy. In the course of a 3-months intervention study the efficacy of a combined protein-rich nutritional therapy with an innovative exercise therapy will be documented for patients with esophageal and bronchial carcinoma in advanced or metastatic stage. An effective stopping of the progress of muscle wasting or even increase of muscle mass, strength and function in the patients of the trial would benefit each patient and his family individually, since it could mean a considerable improvement in his quality of life and tolerability of oncological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal and/or bronchial carcinoma in curative or palliative treatment

Exclusion Criteria:

* Healthy persons or patients under age
* Pregnancy, Lactation
* Psychological disorders, epilepsia, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* Acute cardiovascular disease
* Rheuma
* Intake of anabolic drugs,
* Skin injuries in the area of electrode placements
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Muscle mass maintenance or increase, as assessed by Bioelectrical Impedance Analysis | 12 weeks per patient
  Maintenance or increase of skeletal muscle mass in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS, by assessing Bioelectrical Impedance Analysis values.

SECONDARY OUTCOMES:
Increase in quality of life score by assessing the score points using EORTC-QLQ-C30 questionnaires | 12 weeks per patient
  Clinical improvement by an increase in quality of life in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS.
Increase or maintenance of muscle strength, as assessed by hand grip strength measurements (Jamar dynamometry) | 12 weeks per patient
  Clinical improvement by an increase in muscle strength in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS.
Improvement of pain scores, as assessed by Visual Analog Score | 12 weeks per patient
  Clinical improvement by an increase of pain scores in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS.
Improvement of fatigue scores, as assessed by FACIT-Fatigue Score | 12 weeks per patient
  Clinical improvement by an increase of fatigue scores in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS.
Improvement of oncological therapy tolerance, as assessed by Common Toxicity Criteria regarding gastrointestinal complaints | 12 weeks per patient
  Clinical improvement oncology therapy tolerance in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS.
Maintenance or increase in Body Mass Index (BMI) in kg/m^2-analysis (combination of weight in kilograms and height and in meters | 12 weeks per patient
  Maintenance or increase of skeletal muscle mass in patients with esophagus or bronchial carcinoma receiving a combined therapy of protein-rich nutrition and WB-EMS, by assessing BMI in kg/m^2 (combination of weight in kilograms and height in meters).

CONTACTS AND LOCATIONS:
Overall Officials: Yurdaguel Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- University Hospital Erlangen, Department of Medicine 1, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No